CLINICAL TRIAL: NCT05820061
Title: Pattern Of Endoscopic Findings In Patients Underwent Upper Endoscopy In Sohag University Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aya Ahmed Hassan, resident doctor at Tropical Medicine and Gastroenterology department, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-23-03-04MS
Record Dates: First submitted 2023-03-27; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-03

CONDITIONS: All Patients With Upper GIT Symptoms and Underwent Upper Endoscopy
MeSH Terms: interventions — Gastroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: upper endoscopy — data will be collected from the enoscopy archive files in Department of Tropical Medicine and Gastroenterology,Sohag University Hospital

SUMMARY:
Diseases associated with upper gastrointestinal tract (UGIT) are common and associated with significant morbidity and mortality globally. Peptic ulcer disease, gastroesophageal reflux disease and cancers affect millions of people worldwide.

Upper endoscopy used for various diagnostic and therapeutic utic indications.

DETAILED DESCRIPTION:
Upper GI symptoms are common complaints among the general population and the underlying diseases associated with them carrey significant morbidit.To the best of our knowledge , there is few data about the prevalence rate of various endoscopic findings among Egyptian ptients with UGI symptoms.

Upper gastrointestinal endoscopy (UGIE) is a valuable tool in the diagnosis and management of diseases affecting the esophagus, stomach and upper parts of the duodenum . In addition to direct inspection of the mucosa, endoscopies can be used for therapeutic interventions. Standard diagnostic indications for UGIE include upper gastrointestinal bleeding, evaluation of persistent epigastric pain despite an appropriate trial of therapy, persistent vomiting, dysphagia, anemia, symptoms or signs suggesting structural disease (e.g., anorexia, weight loss,),new onset dyspepsia in a patient older than 50 years of age, heartburn, oesophageal reflux symptoms that persist or recur despite appropriate therapy, surveillance of malignancy, and screening for oesophageal varices in cirrhotic patients. Therapeutic indications include Esophageal variceal ligation, upper GI bleeding control, foreign body removal, dilation or stenting of strictures, placement of feeding tubes, management of achalasia and endoscopic mucosal resection (EMR).

ELIGIBILITY:
Inclusion Criteria: all patients underwent upper endoscopy for various indication at endoscopy unit of Tropical Medicine and Gastroenterology Department, Sohag University Hospital during the specified period of the study

-

Exclusion Criteria:

* Absolute Contraindications

  * Perforated bowel.
  * Peritonitis.
  * Toxic megacolon in an unstable patient. Relative Contraindications
  * Severe neutropenia.
  * Coagulopathy.
  * Severe thrombocytopenia or impaired platelet function.• Increased risk of perforation including connective tissue disorders, recent bowel surgery or bowel obstruction.
  * Aneurysm of the abdominal and iliac aorta

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
spectrum of distribution of endoscopic findings | 2 years
  To assess endoscopic findings in patients presented with upper gastrointestinal symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided